CLINICAL TRIAL: NCT03230123
Title: Effects of Green Banana BIOmass Consumption in Patients With Pre-diabetes and Diabetes MELlitus (The BIOMEL Study)
Acronym: BIOMEL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Maria Cristina de Oliveira Izar, M.D., Ph.D., Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BIO-123
Record Dates: First submitted 2017-07-24; First posted 2017-07-26 (Actual); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Diabetes Mellitus; Pre-diabetes
Keywords: Diabetes Mellitus; green banana; resistant starch; glucose; prebiotics; insulin; incretins
MeSH Terms: conditions — Diabetes Mellitus; Glucose Intolerance; Insulin Resistance

STUDY DESIGN:
Intervention Model Description: Patients with diabetes and Pre-diabetes were randomly allocated to receive diet alone or diet plus green banana biomass suplementation during a six-month intervention period.
Oversight: Data Monitoring Committee: No

ARMS (2):
- Green banana biomass (Experimental): The intervention group is constituted diet counseling plus 4.5 g of resistant starch from green banana biomass, per day, during six months.
  Interventions: Dietary Supplement: Green banana biomass
- Diet alone (Placebo Comparator): The control group will receive diet counseling during six months.
  Interventions: Dietary Supplement: Green banana biomass

INTERVENTIONS:
Dietary Supplement: Green banana biomass — Green banana biomass will be suplemented to diet as 4.5 g per day.

SUMMARY:
Costa ES, Izar MC, Fonseca FAH, França C, Tria H. The benefits of green banana biomass consumption in patients with diabetes mellitus. Federal University of São Paulo, São Paulo, 2015.

According to the Guidelines of the Brazilian Society of Diabetes, Diabetes Mellitus (DM) is a heterogeneous group of metabolic disorders associated with microvascular complications, hyperglycemia, resulting in a higher risk of developing cardiovascular disease. Currently, it is estimated that the world population with diabetes is 382 million people and it is expected to reach 471 million in 2035. About 80% of individuals with diabetes live in developing countries where the epidemic has greater intensity. In the Diabetes Control and Complications Trial and UK Prospective Diabetes Study demonstrated that intensive glycemic control (HbA1c ~ 7.0%) reduces chronic microvascular complications. The resistant starch (RS) is defined as starch and products of its hydrolysis are not absorbed in the small intestine. The green banana presents significant levels of RS, and it is considered a source for the intake of this substance. These foods have physiological functions in the intestinal regulation in glycemic control and delayed gastric emptying. To our knowledge, there are no long-term studies with DM to prove the benefits of resistant starch use. The objective of this study is to assess the benefits of green banana biomass consumption by patients with Pre DM and DM. Considering the possibility of improving glucose, lipid profile, increasing the secretion of glucagon-like peptide-1 (GLP-1), insulin, adiponectin, and reduction in inflammatory markers IL-6, PCR.

DETAILED DESCRIPTION:
INTRODUCTION Cardiovascular Disease and Diabetes In Brazil, chronic non-communicable diseases (NCDs) were the cause of 72% of deaths and reached 63% in the world in 2008, with large numbers of premature deaths. Cardiovascular disease (31.3%), Diabetes Mellitus (DM) (5.2%), cancer (16.3%) and respiratory disease (5.8%) are the main causes of NCDs, leading to loss of quality of life, causing economic impacts that lead to increased poverty. These factors can be reversed through broad interventions and cost-effective health promotion. (Schmidt et al, 2011;. Malta et.al., 2011).

Currently, it is estimated that the world population with diabetes is 382 million people and it is expected to reach 471 million in 2035. About 80% of individuals with diabetes live in developing countries, where the epidemic has greater intensity, with increasing proportion of people affected in younger age groups, coexisting with the problem that infectious diseases still represent. (International Diabetes Federation, 2013; Brazilian Diabetes Society, 2015).

Brazilian data show in 2011 that DM mortality rates (per 100,000 inhabitants) is 30.1 for the general population, 27.2 in men and 32.9 in women, increasing significantly with advancing age, which varies from 0.50 for the age group among 0-29 years to 223.8 for individuals aged from 60 or more, ie an increase of 448 times. (Ministry of Health (USA), 2014; Brazilian Diabetes Society, 2015).

According to the Brazilian Society of Diabetes (2015), DM is a heterogeneous group of metabolic disorders associated to microvascular complications, hyperglycemia, resulting in a higher risk of developing cardiovascular disease (CVD), resulting from defects in insulin action, in insulin secretion or both.

The reference values for diagnosis of DM are glycated hemoglobin (HbA1c)> 6.5% being confirmed in another collecting and dispensable in case of symptoms or glucose> 200 mg and prediabetes HbA1c between 5.7% and 6 4% (Brazilian Society of Diabetes, 2015).

In a meta-analysis carried out with prospective studies it was suggested a significant association of high levels of IL-6 and CRP, with increased risk of diabetes type 2. These results support the hypothesis that chronic inflammation is a predictor of the development of diabetes type 2. IL-6 is a pleiotropic pro-inflammatory cytokine, is produced by a variety of cells including activated leukocytes, endothelial cells and adipocytes. CRP is an acute phase protein plasma and synthesized in the liver. CRP was shown to be a sensitive marker of systemic inflammation (Wang et al., 2013).

The Diabetes Control and Complications Trial (DCCT, 1993) and UK Prospective Diabetes Study (UKPDS, 1998) demonstrated that intensive glycemic control (HbA1c ~ 7.0%) reduces chronic microvascular complications, and can also reduce the occurrence of acute myocardial nonfatal infarction in long term (Ali et al, 2013; American Diabetes Association, 2014; DCCT, 1993; UKPDS, 1998).

In the UKPDS (1998), newly diagnosed type 2 diabetic participants were followed for 10 years and intensive control (mean HbA1c 7.0%) which resulted in reducing the rate of microvascular complications by 25% compared to the conventional treatment (mean HbA1c 7.9%).

The meta-analysis that included three large clinical trials in patients with type 2 diabetes (ADVANCE, ACCORD and VADT) suggests a significant benefit of intensive glycemic control for CVD in participants with newly diagnosed DM, lower HbA1c at baseline and / or in the absence of known CVD (Fonseca et al, 2013;. Skyler, 2009).

The conclusion of the follow-up study of DCCT, that intensive glycemic control started in relatively young individuals, free of CVD risk factors, was associated with a 57% reduction in major CVD, supports the above hypothesis. The DCCT-Epidemiology of Diabetes Interventions and Complications (EDIC) demanded nine years of follow-up after the end of the DCCT, to finally become statistically significant (American Diabetes Association, 2014; DCCT, DTIS, 2008) and demonstrate the effectiveness and benefits in reduce long-term complications of CVD and improve the prospects for a healthy life (DCCT, DTIS, 2014).

Green banana biomass The resistant starch (RS) is defined as starch and products of its hydrolysis are not absorbed in the small intestine. The green banana presents significant levels of RS, and is considered a source for ingestion of this substance (Braga, 2011). These foods have physiological functions in the intestinal regulation, glycemic control, beneficial effects on fatty acid metabolism and delayed gastric emptying. To our knowledge, there are no long-term studies with DM to prove the benefits of resistant starch use (Evert et al., 2014).

The use of RS may reduce the risk of cardiovascular diseases and contributes to weight loss, beyond to promote satiety for a longer period of time (Rahman et al., 2007). The effect of RS on serum lipids in humans are conflicting, however, both studies showed a decrease in total cholesterol and serum triglycerides (Behall, Howe, 1995; Shah, 2012).

The process of digestion and absorption of food takes place primarily in the mammalian intestine, which also releases a group of hormones called incretins. These hormones play an important role in modulating the response of pancreatic islet cells, capable of enhancing insulin secretion, and consequently lead to a decrease of glucagon, thus collaborating to decrease in glucose levels in the blood, especially after meals, when they tend to increase these levels (Doyle, Egan, 2007; Nelson, Cox, 2006).

When the food reaches the intestine, the L and K cells produce GLP-1 and glucose-dependent insulinotropic peptide (GIP), which act in various tissues. In the hypothalamus, they reduce the appetite, sending cholinergic and peptidergic signals to the vagus, inhibiting the antral motility and stimulating the pyloric, thus contributing to the inhibition of gastric emptying. GLP-1 and GIP stimulate the secretion of amylin and insulin and inhibit glucagon release. Insulin has satiating effect on the central nervous system, while amylin slows gastric emptying by vagal action (Tambascia et al., 2014).

Bodinham et al. (2012) examined the effects of the resistant starch consumption on insulin secretion in 12 overweight individuals. The subjects consumed 40 g RS or 27 g of rapidly digestible starch per day for four weeks, separated by a four week washout. The results showed a significant increase in plasma insulin concentrations and C-peptide after four weeks of supplementation with RS compared to placebo. The mechanism of action is unclear, but may be associated with increased secretion of incretins such as GLP-1. On the other hand, Freeland et al. (2010) showed that for occurring increased secretion of GLP-1, the RS intake must be greater than one year. (Bodinham et al., 2014).

One study evaluated 90 subjects with impaired fasting glucose, impaired glucose tolerance or newly diagnosed type 2 diabetes. The intervention group should consume rice containing 6.51 g of RS and the control group should eat rice without supplementation for four weeks. They evaluated the levels of fasting and postprandial glucose and insulin levels, markers of oxidative stress, endothelial function, 24-hour food recall and food frequency questionnaire. The aim of this study was to evaluate whether dietary treatment with rice containing RS for four weeks reduces blood sugar and oxidative stress, as well as promoting the improvement of endothelial function. During the study period, the intervention group showed a tendency to decrease fasting glucose levels, reduction in serum fasting insulin compared to the control group. In patients with impaired fasting glucose, impaired glucose tolerance or newly diagnosed type 2 diabetes in dietary treatment for four weeks with rice containing RS was associated with improvement in endothelial function with a reduction in post-prandial glucose and oxidative stress compared to control group (Kwak et al., 2012).

Bodinham et al. (2014), observed the effect of RS consumption in insulin sensitivity, glucose control and body fat in 17 subjects with type 2 diabetes. The subjects consumed 40 g of RS (derived from corn) or 27 g of a fastly digestible starch per day, during 12 weeks, separated by a washout period of 12 weeks. During the last week of each intervention, participants were instructed to perform the dietary record, bowel habits and symptoms diary, to evaluate the gastrointestinal tolerance of supplements. In the intervention group compared to the control group, increase in triglycerides was observed, but the total cholesterol, adiponectin and leptin showed no change, there was a decrease of TNF and there was no modification in IL-6 and adiponectin, and significantly greater increase in the postprandial GLP-1. The mechanism of action is unclear, but may be associated with increased secretion of incretins (such as GLP-1), which according to the author could act on the muscle for glucose uptake, since there was no change in insulin secretion (Bodinham et al, 2014;. Guimarães et al, 2007)..

Robertson et al. (2012) evaluated 15 men and women with insulin resistance. The intervention included 40 g / day RS derived from corn in comparison to a placebo for eight weeks and eight weeks washout between interventions. There was an increase of glucose uptake in the forearm muscle by analysis arterio - venous forearm muscle (increase of 65% after 15 minutes of RS intake). The function of the adipose tissue was affected with greater suppression of fatty acids after the treatment with RS and an increase in gene expression for the hormone-sensitive lipase, lipoprotein lipase, lipase and fatty triglycerides in the biopsy samples.

Garcia-Rodriguez et al. (2013) evaluated the use of enteral formula for patients with diabetes enriched with RS and the effect on postprandial in 24 healthy or type 2 diabetes subjects. The results showed a lower blood glucose levels in individuals with type 2 diabetes after consumption of enriched formula RS compared to the use of commercially available formulas (Glucerna and Novasource). This indicates that the composition of the enriched formula may have contributed to the improvement of glycemic response after consumption and, therefore, it may have a distinct advantage over the other two classic products. The RS present in the formula can produce a slow, sustained release of glucose into the circulation with a corresponding increase in insulin secretion, which may reduce the risk of hypoglycemia.

Given the above studies of nutritional intervention cited, they were not found long-term, with a considerable sample of individuals with pre-DM and DM and green banana biomass consumption. Thus, it takes long term studies in patients with pre DM and DM to evaluate the benefits of RS consumption, considering the possibility of improved glycemic control, lipid, increase in GLP-1, insulin, adiponectin, and reduction of the inflammation markers IL-6 and CRP.

ELIGIBILITY:
Inclusion Criteria:

* having signed the written informed consent
* males and females aging 18-85 years
* glycated hemoglobin >= 6.5% for diabetic patients
* glycated hemoglobin between 5.7% and 6.4% for pre-diabetic patients
* on stable dose of anti-diabetic drugs and without antecipation of dosage changes during study protocol

Exclusion Criteria:

* use of insulin
* those who need change in dose or addition of medication for diabetes
* any malignancies, except basocelular carcinoma
* heart failure with NYHA class III or IV
* renal failure (GFR< 30 mL/min) or under dialysis therapy
* AIDS
* uncontrolled hypothyroidism (TSH > 10 uUI/mL)
* active liver disease
* severe psychiatric disorders
* any other disease that in the opinion of the investigator could interfere in the results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Percent reduction in glycated hemoglobin | 6 months
  Percent reduction in glycated hemoglobin plasma levels will compare 6 months and baseline levels.

SECONDARY OUTCOMES:
Percent increase in GLP-1 | 6 months
  Percent increase in GLP-1 plasma levels will compare 6 months and baseline levels.

CONTACTS AND LOCATIONS:
Overall Officials: Maria C Izar, M.D., Ph.D., Principal Investigator — Federal University of Sao Paulp
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No